CLINICAL TRIAL: NCT05828875
Title: A Multicenter, Cross-sectional Study on the Quality of Life in Long-term Survival Esophageal Cancer Patients After Radical Radiochemotherapy/Radiotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: bc2022181
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-04

CONDITIONS: Assessing the Current Quality of Life Status of Esophageal Cancer Patients Who Have Undergone Radical Chemoradiotherapy/Radiotherapy and Long-term Survival

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire investigation — Conduct a questionnaire survey on patients' quality of life, nutrition, and psychology

SUMMARY:
This study is a multicenter cross-sectional survey of esophageal cancer patients who underwent radical chemoradiotherapy/radiotherapy from July 2017 to July 2020 in various medical centers, and who survived without disease progression at the time of the survey. The purpose of this study is to evaluate the current quality of life, as well as the incidence of long-term toxic side effects, nutritional status, and psychological status of esophageal cancer patients cured by radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily accept this survey and research;
* The age at the time of radiotherapy is between 18-75 years old, and the age at the time of investigation is<80 years old;
* Histologically confirmed esophageal squamous cell carcinoma without undergoing surgical resection;
* Received radical chemoradiotherapy/radiotherapy from July 2017 to July 2020, currently alive and without disease progression;
* Radiotherapy dose ≥ 45Gy.

Exclusion Criteria:

* Patients who do not cooperate with this survey;
* Patients who have died at the time of investigation;
* Patients who experience tumor progression within the time frame from the end of radiotherapy to receiving this survey;
* Patients diagnosed with other malignant tumors within the time frame from the end of radiotherapy to receiving this survey;
* Patients with incorrect contact information and missing visits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The age at the time of radiotherapy is between 18-75 years old, and the age at the time of investigation is<80 years old;
  * Histologically confirmed esophageal squamous cell carcinoma without undergoing surgical resection;
  * Received radical chemoradiotherapy/radiotherapy from July 2017 to July 2020, currently alive and without disease progression;
  * Radiotherapy dose ≥ 45Gy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Assessment survey | Two years after the end of radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No